CLINICAL TRIAL: NCT04191759
Title: Reliability of the Passive Properties of the Calf Muscles in Healthy Subjects Assessed Using Isokinetic Device
Acronym: ISOSTIFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ISOSTIFF
Record Dates: First submitted 2019-08-27; First posted 2019-12-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2019-12

CONDITIONS: Tendon Injuries; Muscle Tightness
MeSH Terms: conditions — Tendon Injuries

STUDY DESIGN:
Intervention Model Description: One single group of 16 healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test-Retest reproducibility group (Experimental): Protocol is the same for extended or flexed knee. The testing apparatus was set up as described in the constructor owner's manual and subjects were positioned in the supine lying position. The After a 5 min rest period, the participant's ankle is passively stretched through slow loading cycles from 15° of ankle flexion to 35° of ankle extension. Oral instruction is given to the participants to stay relaxed and avoid any muscle contraction and movement of the leg throughout the passive stretching. To familiarize, participant have 3 repetitions of passive ankle flexion-extension at 5°.s-1, and after 2min rest, data are collected from one repetitions at 5°.s-1 in passive mode. The measurements are also performed at an angular rate of 90°.s-1, according to the same protocol. Data for maximal voluntary isokinetic contraction are collected from 3 maximal repetitions at 60°.s-1 in concentric mode and participant are encouraged by constant verbal stimulation.
  Interventions: Diagnostic Test: Test-Retest reproducibility

INTERVENTIONS:
Diagnostic Test: Test-Retest reproducibility — Protocol is the same for extended or flexed knee. The testing apparatus was set up as described in the constructor owner's manual and subjects were positioned in the supine lying position. The After a 5 min rest period, the participant's ankle is passively stretched through slow loading cycles from 15° of ankle flexion to 35° of ankle extension. Oral instruction is given to the participants to stay relaxed and avoid any muscle contraction and movement of the leg throughout the passive stretching. To familiarize, participant have 3 repetitions of passive ankle flexion-extension at 5°.s-1, and after 2min rest, data are collected from one repetitions at 5°.s-1 in passive mode. The measurements are also performed at an angular rate of 90°.s-1, according to the same protocol. Data for maximal voluntary isokinetic contraction are collected from 3 maximal repetitions at 60°.s-1 in concentric mode and participant are encouraged by constant verbal stimulation.

SUMMARY:
The investigators designed this study to determine the test-retest reliability of the viscoelastic passive properties of the calf muscles assessed using isokinetic device in flexed and extended knee position. The second objective is to determine the clinical viability of the parameters using the coefficient of repeatability and to investigate the individual characteristics associated with increased calf stiffness or altered viscoelasticity

DETAILED DESCRIPTION:
Recordings using an isokinetic dynamometer make it possible to quantify the resisting force during passive muscle stretch for a constant speed movement in dorsal flexion (flexion) and its release in plantar flexion (extension). The surface electromyography (EMG) makes it possible to measure voluntary contraction and the movement is considered passive if the corrected and normalized EMG signal, using root-mean-square (RMS), is less than 10% RMS during the Maximal Voluntary Muscle Contraction (MVMC).

Stiffness is calculated from the slope of the rise of the curve during the passive dorsiflexion phase of the joint. The elastic potential energy can be measured and corresponds to the area under the curve during elongation.

During the plantar flexion return phase, there is a hysteresis phenomenon resulting in behavior that differs from the curve. This difference between the two curves corresponds to the behavior related to viscoelastic relaxation. Viscoelasticity has a thixotropic behavior, i.e. it varies over time, for example, with heating. These parameters have been studied together or separately to evaluate the effect of age or stretching on the passive mechanical properties of the calf.

However, the test-retest reliability of the viscoelastic passive properties of the calf muscles assessed using isokinetic device has not been demonstrated.

The investigators designed this study to determine the test-retest reliability of the viscoelastic passive properties of the calf muscles assessed using isokinetic device in flexed and extended knee position. The second objective is to determine the clinical viability of the parameters using the coefficient of repeatability and to investigate the individual characteristics associated with increased calf stiffness or altered viscoelasticity

Muscle tension is expressed by the peak torque (Nm), recorded at neutral position (PT0°) and 10° flexion (PT10°). Plantarflexor stiffness is determined as the slope of the torque-angle curve expressed as Nm·degree-1 during the linear region form 0-10° flexion (Slope0-10). A measure of elastic energy storage is calculated through the AUC of the torque-angle curve across the all range of motion. Hystérésis over time due to viscoelastic stress relaxation is calculated as the percent reduction in work absorption between the muscle stretching and releasing phases . The flexed-to-extended ratio is calculated as the ratio of flexed knee to extended knee and evaluated for PT0°, PT10° and Slope0-10 values , at 5 and 90°/sec

ELIGIBILITY:
Inclusion Criteria:

* Patient who signed the research information form
* Patient affiliated to a social security system
* An active patient, under 45 years of age, who participates in at least 4 hours of physical activity per week

Exclusion Criteria:

* Individuals unable to perform an isokinetic muscle testing
* Individuals with a current or recent lower limb injury with time loss from sport participation within the previous month.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline stiffness parameters at 15 days to assess the reproducibility of stiffness parameters | Two evaluations on both dominant and non dominant knees: one evaluation at the first visit, and a second evaluation at the second visit at 15 days after the first visit
  Change from Baseline stiffness parameters at 15 days, measurement of passive peak torque at 0 and 10° and slope of curve during the passive ankle flexion using an isokinetic device
Change from Baseline viscoelastic parameters at 15 days to assess the reproducibility of viscoelastic parameters | Two evaluations on both dominant and non dominant knees: one evaluation at the first visit, and a second evaluation at the second visit at 15 days after the first visit
  Change from Baseline viscoelasticity parameters at 15 days, measurement of hysterisis (AUC release/AUC storage) during the passive ankle flexion/extension using an isokinetic device

SECONDARY OUTCOMES:
Patient characteristics | One evaluation only, at the first visit after inclusion
  Personal characteristics recorded in the medical report as age, gender, type of sport and sport level of practice and previous lower limb injuries
Physical characteristics, popliteal angle | One evaluation only, at the first visit after inclusion
  The popliteal angle tested on both legs.
Physical characteristics, Calf Circumference | One evaluationsonly, at the first visit after inclusion (T1)
  The Calf Circumference (CC) tested on both legs.
Physical characteristics, ROM | One evaluation only, at the first visit after inclusion
  The passive ankle range of motion (ROM) tested on both legs.
Physical characteristics, Fingertip-to-Floor (FTF) Test | One evaluation only, at the first visit after inclusion
  The Fingertip-to-Floor (FTF) Test on both legs.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided